CLINICAL TRIAL: NCT07143253
Title: Evaluation of 1-year Survival Rates of Two Different Fissure Sealants Applied to Immature Permanent Molars
Brief Title: One-year Survival of Fissure Sealants in Immature Permanent Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Handan Vural (Other)
Responsible Party: Sponsor-Investigator, Handan Vural, assistant professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 7699
Record Dates: First submitted 2025-08-10; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Evaluation of the Survival of Different Fissure Sealants in Partially Erupted Immature Molar Teeth at Various Eruption Stages
Keywords: immature molars; Fissure Sealant; Partially Erupted

STUDY DESIGN:
Intervention Model Description: In this split-mouth designed study, at least two partially erupted molar teeth from each patient will be included. A random group allocation will be performed, and the appropriate fissure sealant will be applied according to the assigned group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gruop A:UltraSeal XT hydro sealant / hydrophillic pit and fissure sealent (Active Comparator): The presence of moisture and saliva-contamination during the placement of the sealant compromise the quality of adhesion at the sealant-enamel interface, which impacts the ongoing resistance to microleakage of microorganisms. Hydrophilic sealants, which bond effectively to moist enamel surfaces, present a distinct advantage in paediatric dentistry where patient-compliance, isolation, and moisture-control can be particularly challenging.UltraSeal XT® hydro™ is a new moisture-tolerant, self-adhesive, light-cured, acrylate-based, hydrophilic pit, and fissure sealant which has been developed by Ultradent Products, USA. The sealant comprises a 53 wt% mixture of inorganic filler particles that confer radiopacity. This material is reported to "chase" moisture into the pits and fissures, thus eliminating moisture-related failure associated with hydrophobic sealants
  Interventions: Procedure: Preventive pit and fissure sealant application
- Gruop B: GC Fuji Triage- glassionomer pit and fissure sealent (Active Comparator): Glass ionomer (GI)-based fissure sealants are considered a valuable treatment alternative, particularly in pediatric dentistry for patients at high risk of caries, due to their ability to chemically bond to dental tissues, release fluoride, exhibit biocompatibility, provide antibacterial effects, and promote the remineralization of hydroxyapatite crystals. The self-bonding, high-fluoride-releasing GC Fuji TRIAGE® is frequently reported in the literature as a fissure sealant, particularly for immature and partially erupted teeth. The use of glass ionomers as fissure sealants is especially emphasized in cases where isolation is difficult.
  Interventions: Procedure: Preventive pit and fissure sealant application

INTERVENTIONS:
Procedure: Preventive pit and fissure sealant application — Preventive pit and fissure sealant application is a preventive procedure involving the use of flowable resin-based or glass ionomer-based materials to physically cover the occlusal surfaces of teeth, particularly in pits and fissures at high risk of caries development. This barrier prevents plaque accumulation and protects the enamel surface.
  In this study, no procedures beyond the routine clinical application of the materials will be performed. However, partially erupted permanent teeth with challenging isolation will be specifically selected. Both materials will be applied using a split-mouth design to the teeth of the same participant. This approach will allow for an effective and comparative evaluation of the clinical retention of the material.

SUMMARY:
Dental caries remains one of the most prevalent oral diseases today. The risk of caries development is highest during the first few years following tooth eruption. Therefore, preventive strategies for dental caries continue to be of great importance.

In particular, permanent second molars are highly susceptible to caries during their eruption phase, as the enamel has not yet completed its physiological maturation. This vulnerability is especially pronounced in partially erupted teeth, where the risk of caries formation increases significantly in the absence of effective preventive measures.

In this context, fissure sealants are widely used as a preventive approach, particularly in children and adolescents, due to their proven efficacy in caries prevention. In this study, the 12-month clinical performance of resin-based hydrophilic and glass ionomer-based fissure sealants applied to partially erupted permanent first and/or second molars will be evaluated comparatively.

Informed consent will be obtained from all participants prior to their inclusion in the study. The aim of this research is to provide scientific evidence to support material selection in the field of preventive dentistry.

Previous studies (Ahovuo-Saloranta et al., 2013) have emphasized that long-term clinical success rates have a direct impact on material selection, highlighting the importance of conducting prospective clinical trials.

This study is designed as a split-mouth, double-blind, randomized, controlled clinical trial. The reporting of the study will adhere to the CONSORT (Consolidated Standards of Reporting Trials) guidelines. The study will be conducted at the Department of Pediatric Dentistry, Faculty of Dentistry, İnönü University.

Healthy children aged between 7 and 15 years will be included in the study. Randomization will be performed using a computer-assisted program. Two different fissure sealants will be applied to different teeth in each patient.

Application Procedure:

All fissure sealants will be applied by a single experienced operator in accordance with the manufacturer's instructions.

Resin-based sealants will be polymerized for 20 seconds using an LED light source.

Group A: Hydrophilic fissure sealant

Group B: Glass ionomer-based fissure sealant

Evaluation Time Points:

Immediately after application

At 3 months

At 6 months

At 12 months

The following parameters will be assessed by two independent blinded evaluators according to modified USPHS criteria:

Retention of the fissure sealant (Complete / Partial / Total loss)

Marginal discoloration

Development of secondary caries

Data will be entered into Microsoft Excel and analyzed using SPSS software. A p-value of < 0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
This study is designed to compare the 12-month survival rates of GC Fuji Triage (glass ionomer-based) and UltraSeal XT™ hydro™ (Hydrophilic Pit and Fissure Sealant) fissure sealants applied to partially erupted permanent second molars. The research will be conducted using a split-mouth, double-blind, randomized, and controlled design, aiming to provide a high level of scientific reliability through its prospective nature.

Blinding of both participants and evaluators is intended to minimize observational bias and enhance the validity of the results. The study is expected to provide evidence-based data that will guide clinicians in material selection and contribute to the existing literature in the field.

Furthermore, by being reported in accordance with the CONSORT guidelines, the study will meet international standards for clinical research reporting.

Inclusion Criteria:

Healthy children aged 10 to 15 years. Partially erupted, caries-free or demineralized fissures with ICDAS scores 1-2 on permanent second molars, confirmed by clinical and radiographic examination.

Children who demonstrate cooperative behavior, scoring 3 or 4 on the Frankl Behavior Rating Scale.

An oral hygiene score (OHI-S) ≤ 3. Written informed consent obtained from a parent or legal guardian prior to participation in the study.

Exclusion Criteria:

Fully erupted or completely impacted teeth. Teeth with severe hypoplasia, hypomineralization, presence of extensive restorations, or cavitated carious lesions.

Children with a history of systemic disease or long-term medication use. Known allergies to resin-based or glass ionomer materials. Presence of parafunctional habits (e.g., bruxism, nail biting, etc.).

Two different fissure sealants will be applied to different teeth in each patient.

Application Procedure:

All fissure sealants will be applied by a single experienced operator in accordance with the manufacturer's instructions.

Resin-based sealants will be light-cured for 20 seconds using an LED curing light.

Group A: Hydrophilic fissure sealant

Group B: Glass ionomer-based fissure sealant

Evaluation Time Points:

Immediately after application At 3 months At 6 months At 12 months

The following parameters will be evaluated by two independent blinded evaluators according to modified USPHS criteria:

Sealant retention (Complete / Partial / Total loss) Marginal discoloration Development of secondary caries

In cases where sealant loss is observed during follow-up, the material will be reapplied to the affected tooth; however, that tooth will not be included in subsequent evaluations.

Participants will not experience any disadvantage or harm due to any adverse outcome related to the materials used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 10-15 years.
* Partially erupted second permanent molars that are clinically and radiographically confirmed to be caries-free or present with demineralized fissures scored as ICDAS 1-2.
* Children demonstrating cooperative behavior, with a Frankl Behavior Rating Scale score of 3 or 4.
* Oral Hygiene Index (OHI-S) score ≤ 3
* Written informed consent obtained from the parent or legal guardian.

Exclusion Criteria:

* Fully erupted or completely impacted teeth.
* Teeth presenting with severe hypoplasia, hypomineralization, extensive restorations, or cavitated carious lesions.
* History of systemic disease or long-term medication use.
* Known allergy to resin-based or glass ionomer materials.
* Presence of parafunctional habits.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Modified Simonsen Criteria | Follow-up appointments were scheduled for children at 3, 6, and 12 months following the initial treatment.
  Score 0 Fissure sealant is completely in the mouth and there is no new caries.
  Score 1 Partial loss of fissure sealant, no new caries.
  Score 2 Partial loss of fissure sealant and new caries.
  Score 3 Complete loss of fissure sealant, no new caries.
  Score 4 Complete loss of fissure sealant and new caries
Edge Integrity Evaluation Criteria | Follow-up appointments were scheduled for children at 3, 6, and 12 months following the initial treatment
  0: The fissure sealant and tooth surface are intact and cannot be distinguished with a probe.
  1. The edges of the fissure sealants can be distinguished with a probe.
  2. There is a gap along the edge of the fissure sealant and deep cracks reaching the central fossa
Marginal Coloration Evaluation Criteria | Follow-up appointments were scheduled for children at 3, 6, and 12 months following the initial treatment
  0 No color change between fissure sealant and tooth.
  1. Color change in only one area.
  2. Color change in many areas.
  3. Severe color change indicating leakage.
Anatomical Form Evaluation Criteria | Follow-up appointments were scheduled for children at 3, 6, and 12 months following the initial treatment.
  0 Consistent with and continuous with occlusal form and structure.
  1. Change in anatomical form but all pits and fissures covered.
  2. a Partial loss of one or two pits or fissures but no need to repair or replace fissure sealant.
  2b Partial loss of pits and fissures, fissure sealant needs to be replaced or repaired.
  3 Loss of all pits and fissures. 7 Partial loss due to occlusion 9 Bleb not connected to margins

CONTACTS AND LOCATIONS:
Overall Officials: handan vural, Assistant Professor, Study Chair — Department of Pediatric Dentistry, Faculty of Dentistry, Inonu University
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dentistry, Inonu University, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 6 months and ending 1 years after the publication of results"
Access Criteria: Access to individual participant data (IPD) and supporting materials will be made available to qualified researchers upon reasonable request. The following details apply:
  Who can access the data: Qualified academic researchers with a valid scientific purpose.
  What can be accessed: De-identified IPD, study protocol, statistical analysis plan, informed consent forms, and ethics approval documents.
  How to access: Interested researchers must submit a written request, including a brief research proposal and documentation of ethics committee approval. Requests should be sent to the corresponding author via email. Data sharing will be conducted in accordance with ethical guidelines and applicable data protection regulations.

REFERENCES:
- [Background] Penha KJS, Roma FRVO, Filho EMM, Ribeiro CCC, Firoozmand LM. Bioactive self-etching sealant on newly erupted molars: A split-mouth clinical trial. J Dent. 2021 Dec;115:103857. doi: 10.1016/j.jdent.2021.103857. Epub 2021 Oct 24. PMID 34699954
- [Background] Antonson SA, Antonson DE, Brener S, Crutchfield J, Larumbe J, Michaud C, Yazici AR, Hardigan PC, Alempour S, Evans D, Ocanto R. Twenty-four month clinical evaluation of fissure sealants on partially erupted permanent first molars: glass ionomer versus resin-based sealant. J Am Dent Assoc. 2012 Feb;143(2):115-22. doi: 10.14219/jada.archive.2012.0121. Erratum In: J Am Dent Assoc. 2012 Apr;143(4):336. PMID 22298552